CLINICAL TRIAL: NCT04938128
Title: The Effect of CPAP on Nocturnal Dipping in Normotensive Patients With Moderate-severe Obstructive Sleep Apnoea, a Multicentre Randomised Controlled Trial
Brief Title: Effect of CPAP vs Control on Nocturnal Dipping in Normotensive Patients With Obstructive Sleep Apnea
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit
Sponsor: St Vincent's University Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Dr Silke Ryan, Clinical Professor, Consultant in Respiratory and Sleep Medicine, St Vincent's University Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RS21-008
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Continuous positive airway pressure; Non-dipper; Normotensive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP treatment (Experimental): This group will receive CPAP treatment
  Interventions: Device: CPAP
- Control (No Intervention): This group will receive Diet and Lifestyle advice only

INTERVENTIONS:
Device: CPAP — Gold standard treatment for obstructive sleep apnea. In this group, patients will be prescribed CPAP treatment according to local policy.
  Arms: CPAP treatment

SUMMARY:
This is an open-label, parallel, prospective, randomised control trial evaluating the effect of Continuous Positive airway pressure (CPAP), the standard treatment for obstructive sleep apnea (OSA) versus control (diet and lifestyle advice) on dipping status and blood pressure parameters in 100 non-dipper normotensive patients with moderate to severe obstructive sleep apnea and without established cardiovascular or metabolic disease.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed moderate-severe OSA (by standard criteria)
* Absence of known hypertension and antihypertensive medication
* Office blood pressure <140/90mmHg
* Age 18 - 70 years
* Able to provide written, informed consent

Exclusion Criteria:

* Pregnancy
* Previous diagnosis of OSA or previous CPAP treatment
* Diagnosis of Diabetes Mellitus
* Active treatment for malignancy or severe psychiatric disorder
* History of cardiovascular disease or cerebrovascular disease
* Moderate or severe chronic kidney disease (CKD) defined as a eGFR of ≤ 44mL/min/1.73m2
* Dipper on ABPM
* Morbid obesity, defined as BMI ≥40
* Professional drivers or drivers with a history of road-traffic accident due to sleepiness
* Severe excessive daytime sleepiness defined as Epworth sleepiness scale (ESS) >15

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Dipping status | 3 months
  Change in % dipping after 3 months of treatment with CPAP versus Control

SECONDARY OUTCOMES:
Change in the mean 24-hour ambulatory blood pressure (BP) | 3 months
  Change in mmHg in mean blood pressure from baseline to 12 weeks of treatment compared to control
Change in blood pressure parameters | 3 months
  Change in mmHg in blood pressure parameters including diurnal and nocturnal systolic blood pressure (SBP) and diastolic blood pressure (DBP) from baseline to 12 weeks of treatment compared to control

CONTACTS AND LOCATIONS:
Locations (1):
- St Vincent's University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No